CLINICAL TRIAL: NCT03682991
Title: Reversal of Atrial Substrate to Prevent Atrial Fibrillation
Brief Title: Reversal of Atrial Substrate to Prevent Atrial
Acronym: RASTA AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Abbott (Industry); Phillips (Unknown); Cardiac Arrhythmia Network of Canada (Other)
Responsible Party: Principal Investigator, Ratika Parkash, Attending Staff, Department of Medicine, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP-007
Record Dates: First submitted 2018-08-27; First posted 2018-09-25 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This will be a parallel group, open label randomized clinical trial, with blinded endpoint evaluation (PROBE design)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aggressive Risk Factor Control (Experimental): Multifaceted risk factor management relating to BP, exercise, sleep apnea, alcohol intake and diabetes management
  Interventions: Other: Aggressive Risk Factor Control
- Standard of Care (Active Comparator): All patients in the control arm will receive therapies for AF as per the existing guidelines. BP, cholesterol, diabetic management will be administered as per the available guidelines.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Aggressive Risk Factor Control — 1. Sleep apnea screening, therapy is recommended if apopnea-hypopnea (AHI) index is greater than 15, with a target index of less than 5.
  2. Counseling regarding alcohol reduction to 2 drinks/day for men, 1 drink/day for women, no binge drinking (>5 drinks at one setting).
  3. Participation in a 12 week structured, home-based exercise program and nutritional counseling. Weight reduction will be emphasized through modification of diet and exercise.
  4. Blood Pressure management to achieve a target systolic blood pressure (SBP) of <120/80 mm/Hg
  5. Smoking cessation facilitated through local resources already established at each site
  Arms: Aggressive Risk Factor Control
Other: Standard of Care — Recommendations based on current guidelines
  Arms: Standard of Care

SUMMARY:
A multi-center, randomized trial to examine the effect of aggressive risk factor control and arrhythmia trigger-based intervention on recurrence of atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a major health problem, with a prevalence of 0.4-1% of the population. It results in high healthcare costs and significant morbidity, especially for patients with severe symptoms. Exercise and risk factor modification to prevent and modify AF has garnered a significant amount of support in cohort studies that have proven benefit. It is well known that age, body mass index, valvular heart disease, heart failure, hypertension and sleep apnea are risk factors for AF, most of which are modifiable if targeted appropriately. In addition, catheter ablation techniques have evolved and improved to reduce AF recurrence in those who are most symptomatic, and either have heart failure, or are at risk for its development. Despite these advances, the recurrence of AF remains high.

We propose to determine whether early treatment of the arrhythmogenic substrate, with or without aggressive risk factor modification, is most important in prevention of recurrent AF. It is hypothesized that patients with underlying risk factors that promote AF will benefit most from a combined strategy of aggressive risk factor modification in combination with catheter ablation.

The study design will be a two-arm, parallel group, randomized clinical trial comparing catheter ablation versus catheter ablation plus aggressive risk factor therapy, followed by maintenance with blinded endpoint evaluation. Patients with symptomatic AF and two of the following will be included: BP ≥ 140/90 or history of hypertension, BMI≥27, diabetes, prior stroke/TIA, history of heart failure (prior heart failure admission due to AF or LVEF<40%), age≥65. Patients will be excluded if they are exercising >150 minutes/week by self-report. Patients will be randomly allocated to one of the following groups: 1) AF ablation within 3 months, 2) AF ablation at 3 months, with a 12 week home-based exercise/risk factor management program, followed by maintenance therapy. A 5-month treatment period will be observed to deliver the interventions and have a 2 month blanking period post ablation. Guideline-directed therapy for risk factors will occur in all groups, including BP, cholesterol, diabetes, alcohol reduction and sleep apnea screening. All patients will undergo implantation of an implantable cardiac monitor (ICM) at baseline. The primary outcome will be a composite of clincally significant AF (AF ≥ 24 hours), AF-related hospitalization/emergency department visits 5 months post randomization. Secondary outcomes will include: Death, Stroke or Systemic embolism, Quality of Life, Health Outcomes, recurrent AF, & AF burden. The sample size required is 500. Safety outcomes include: AF catheter ablation procedural complications, Anti-arrhythmic medication related adverse events, & Death.

ELIGIBILITY:
Inclusion Criteria: Patients with symptomatic (CCS-SAF ≥2) paroxysmal or persistent atrial fibrillation despite rate control, desiring catheter ablation and at least two of the following:

* BMI ≥ 27,
* BP ≥140/90 mmHg or history of hypertension,
* Prior stroke/transient ischemic attack,
* Diabetes,
* Heart failure (prior heart failure admission or left ventricle ejection fraction (LVEF) <40%),
* Age ≥ 65 years
* Current smoker
* Excessive Alcohol use

Exclusion Criteria:

* Permanent AF (AF lasting > 3 years)
* Prior catheter ablation for AF
* New York Heart Association (NYHA) Class IV (Severe) heart failure,
* Participation in a cardiac rehabilitation program within the last year,
* Currently performing exercise training >150 minutes/week of moderate to vigorous physical activity,
* Unable to exercise,
* Unable to give informed consent,
* Other noncardiovascular medical condition making 1 year survival unlikely,
* Less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of AF related hospitalizations post ablation | up to 72 months
  AF-related hospitalizations (lasting more than 24 hours) from 2-months post ablation to end of follow up.
Number of AF related Emergency Department (ED) visits post ablation | up to 72 months
  AF-related emergency department visits from 2-months post ablation to end of follow up.
Number of clinically significant AF events post ablation | up to 72 months
  Clinically significant AF events lasting >24 hours (either an irregular R-R interval, or atrial cycle length < 280 ms, as obtained from an insertable cardiac monitor) from 2-months post ablation to end of follow up.

SECONDARY OUTCOMES:
Number of AF-related hospitalizations | up to 72 months
  AF-related hospitalizations (lasting more than 24 hours) from randomization to end of follow up.
Number of AF-related emergency department (ED) visits | up to 72 months
  AF-related emergency department visits from randomization to end of follow up.
Number of Clinically significant AF events | up to 72 months
  Clinically significant AF events lasting >24 hours (either an irregular R-R interval, or atrial cycle length < 280 ms, as obtained from an insertable cardiac monitor) from randomization to end of follow up.
Mean AF burden | up to 72 months
  Average percentage of time in AF during follow up, as measured by insertable cardiac monitor.
Stroke or systemic embolism events | up to 72 months
  Total number of stoke or systemic embolism events.
Quality of Life - CCS-SAF | Up to 24 months
  Symptom burden as measured by the Canadian Cardiovascular Society (CCS) Severity of Atrial Fibrillation (SAF) scale. CCS-SAF scores range from 0 to 4, with higher values representing more severe impact of symptoms on quality of life and activities of daily living.
Quality of Life - AFEQT | Up to 24 months
  Quality of life as measured by the Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) scale. The scale consists of 21 questions with 7-point Likert scale responses. Questions 1-18 are grouped into three subscales (symptoms, daily activities and treatment concern). Questions 19-21 capture satisfaction with treatment and are not include in the HRQoL score of the questionnaire. Overall and subscale scores range from 0 to 100. Lower scores correspond to higher levels of disability (e.g., 0 corresponds to complete disability or responding "extremely" limited, difficult or bothersome to all questions answered), while a score of 100 corresponds to no disability (e.g., responding "not at all" limited, difficult or bothersome to all questions answered). For Satisfaction questions, a score of 100 corresponds to extreme satisfaction with current treatment.
Number of recurrent AF-ablations | up to 72 months
  Number of re-ablations required.
Cardioversions | up to 72 months
  Number of cardioversions required.
All-cause mortality | up to 72 months
  Any deaths occurring at any time during the study.
AF at any time | Up to 72 months post randomization
  Atrial fibrillation (confirmed by ICM, 12-lead ECG or telemetry)
Health Outcomes | Up to 24 months
  Measured by the Euroqol-5D-5L questionnaire
Association between gender, AF risk factors and aggressive risk factor management | UP to 24 months
  This will be determined by the use of the GENESIS Praxy Gender questionnaire
Major Bleeding | Up to 72 months
  Any event which includes the following criteria: fall in Hgb of ≥2 g/dL, transfusion of ≥2 units PRBC or whole blood, in a critical location (e.g., intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial), causes death

OTHER OUTCOMES:
Number of ablation procedural complications [Safety] | up to 72 months
  Periprocedural complications will be assessed.
Number of antiarrhythmic drug adverse effects [Safety] | up to 72 months
  Adverse drug reactions will be assessed.
Death (Safety) | Up to 72 months
  All cause mortality occurring at any time post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Ratika Parkash, Principal Investigator — Nova Scotia Health Authority; Allan Skanes, Study Director — London Health Sciences Centre; Chris Blanchard, Study Director — Nova Scotia Health; David Birnie, Study Director — University of Ottawa Heart Institution; George Wells, Study Director — University of Ottawa Heart Institution; Michiel Rienstra, Study Director — University of Groningen; Jeff Healey, Study Director — Hamilton Health Sciences Centre; Jennifer Reed, Study Director — University of Ottawa Heart Institution; Anthony Tang, Study Director — London Health Sciences Centre; Vidal Essebag, Study Director — McGill University Hospital; Isabelle vanGelder, Study Director — University of Groningen; John Sapp, Study Director — Nova Scotia Health Authority
Locations (17):
- Canada (17):
  - Foothills Hospital, Calgary, Alberta
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - Kelowna General Health, Kelowna, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Center, Hamilton, Ontario
  - St. Mary's General Hospital, Kitchener, Ontario
  - London Health Sciences Center, London, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Laval Hospital, Laval, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Sacre Coeur Hospital, Montreal, Quebec
  - Regina General Hospital, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No